CLINICAL TRIAL: NCT05841862
Title: Intravitreal Quantum Dots (QD) for Advanced Retinitis Pigmentosa (QUANTUM): a Pilot, Randomized, Double-masked, Sham-controlled, Clinical Device Trial
Brief Title: Intravitreal Quantum Dots (QD) for Advanced Retinitis Pigmentosa (RP) (QUANTUM)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding.
Sponsor: 2C Tech Corp (Industry)
Collaborators: ORA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2C Tech-002
Record Dates: First submitted 2023-04-24; First posted 2023-05-03 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2024-12

CONDITIONS: Retinitis Pigmentosa
MeSH Terms: conditions — Retinitis Pigmentosa

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be masked to the assignment of which eye is receiving active treatment or sham treatment. Clinical personnel who perform clinical assessments will also be masked to the participants' eye assignment. Masked evaluators will not be permitted in the room during the injections and will be instructed to avoid areas where they may observe study activities which may potentially lead to their becoming unmasked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 2C-QD (Experimental): Single-dose intravitreal injection
  Interventions: Device: 2C-QD
- Sham 2C-QD (Sham Comparator): Single-dose intravitreal injection
  Interventions: Device: Sham 2C-QD

INTERVENTIONS:
Device: 2C-QD — Quantum Dot
  Arms: 2C-QD
Device: Sham 2C-QD — Sham Intravitreal Injection
  Arms: Sham 2C-QD

SUMMARY:
Pilot, randomized, observer and participant masked, sham and fellow eye controlled, interventional clinical device trail to evaluate the safety and effectiveness of the 2C-QD device to improve visual function in adults with advanced Retinitis Pigmentosa (RP).

DETAILED DESCRIPTION:
Subjects will be informed about the study and potential risks and benefits, and then will provide written informed consent prior to study procedures being performed. Subjects will be screened for eligibility against criteria set forth within the clinical protocol. If subjects are eligible, they will be randomized to receive an intravitreal injection of the 2C-QD device in one eye, and the fellow eye will receive a sham injection and serve as the control. Subjects will then be following for 180 days, through 9 visits.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female adults, aged 18 years or older on the day of screening
2. Clinical diagnosis of bilateral RP, based on two or more of the following: clinical features, visual field testing, retinal imaging, electrophysiological measures, or genetic testing
3. BCVA of 6/60 (logMAR 1.0) or worse in both eyes, with loss of vision due to RP in the opinion of the Investigator.
4. Central visual field of less than 20 degrees in both eyes
5. Be able to follow instructions and ambulate
6. Be able to complete at least one mobility course at highest luminance level using each eye separately
7. Be able and willing to provide written informed consent, attend all scheduled visits and comply with all study procedures
8. For females capable of becoming pregnant, agree to have urine pregnancy testing (must be negative) and must not be lactating; and must agree to use a medically acceptable form of birth control throughout the study duration. Women considered capable of becoming pregnant include all females who have experienced menarche and have not experienced menopause (as defined by amenorrhea for greater than 12 consecutive months) or have not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy). Acceptable forms of birth control are spermicide with barrier, oral contraceptive, injectable or implantable method of contraception, transdermal contraceptive, intrauterine device, or surgical sterilization of partner. For non-sexually active females, abstinence will be considered an acceptable form of birth control.

Exclusion Criteria:

1. Presence of severe systemic disease resulting in a life expectancy shorter than 1 year
2. Presence of retinal or optic nerve disease other than RP in either eye including cystoid macular oedema (CMO), glaucoma or ocular hypertension (IOP≥ 25mmHg), diabetic retinopathy, retinal vein occlusion, and age-related macular degeneration.
3. Be currently using any topical therapy for CMO (e.g., carbonic anhydrase inhibitors, corticosteroids, NSAIDs) in either eye.
4. Have the presence of an ocular media opacity in either eye, which in the opinion of the Investigator, will preclude an accurate evaluation at any time during the study
5. Have the presence of active ocular or systemic infection or inflammation, or any history of intraocular inflammation in either eye
6. Have had a prior vitrectomy in either eye
7. Have a history of amblyopia in either eye
8. Have current or former high myopia (>6 dioptres) in either eye
9. Have undergone ocular surgery within 6 months of the screening visit in either eye or have planned ocular surgery in either eye
10. Have one eye that is ineligible, or have asymmetrical ocular disease defined as a greater than 15 letter difference between the eyes based on BCVA results.
11. Have participated in any study involving an investigational drug or device within the past 30 days or have ongoing participation in a study with an investigational drug or device or have participated in a clinical trial of gene or cell therapy at any time
12. Have any clinical evidence that the Investigator feels would place the subject at increased risk with the investigational product

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-03-20 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Monocular navigation performance | baseline to week 2
  measured based on the ability to navigate the course under different light levels (defined as luminance) using the mobility course.

SECONDARY OUTCOMES:
Monocular navigation performance | baseline to week 4, 12, 24, 52
  measured using luminance level to complete the mobility course
binocular navigation performance | baseline to week 2, 4, 12, 24, 52
  measured using luminance level to complete the mobility course
monocular retinal sensitivity | baseline to week 2, 4, 12, 24, 52
  measured using Octopus full-field static perimetry
monocular best-corrected visual acuity (BCVA) | baseline to week 2, 4, 12, 24, 52
  change in BCVA
ellipsoid zone area | baseline to week 2, 4, 12, 24, 52
  measured using spectral domain (SD) optical coherence tomography (OCT)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Jackson, Professor, Principal Investigator — Kings College Hospital

IPD SHARING:
Plan to Share IPD: No